CLINICAL TRIAL: NCT05627349
Title: The Evaluation for Fu's Subcutaneous Needling in Carpal Tunnel Syndrome: a Randomized Controlled Trial.
Brief Title: The Evaluation for Fu's Subcutaneous Needling (FSN) in Carpal Tunnel Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH111-REC2-065
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Fu's Subcutaneous Needling, carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wrist splinting group (Experimental): wrist splinting at night for 2 weeks
  Interventions: Device: wrist splinting
- FSN group (Experimental): The needle inserted at the midpoint of the anterior forearm of the affected side. Swaying movement (SM) frequency is 200 times in 2 minutes. Reperfusion approach (RA) was performed with slow repetitively grasping movement while SM. On the 1st, 2nd, and 4th days, three times of FSN treatment were arranged.
  Interventions: Device: FSN

INTERVENTIONS:
Device: wrist splinting — standard wrist splinting at night for 2 weeks
  Arms: wrist splinting group
Device: FSN — FSN is a single-use disposable needle(Trocar Acupuncture Needle, Nanjing FSN Medical Co. , Ltd, China.). The needle body is solid, and covered with a plastic tube. The needle penetrates the skin with insertion device. Under the guidance of ultrasound, the needle enter the loose subcutaneous layer obliquely without penetrating into the muscle. This is the difference from traditional acupuncture. The insertion point is midpoint of the anterior forearm. The needle tip is toward the carpal tunnel. After the needle is inserted, SM and RA are performed. The frequency of SM is 200 times in two minutes. The method of SM is to make a horizontal fan swaying with the base of the needle as the fulcrum. RA is performed while SM-slowly make a fist for 10 seconds and then relax for 5 seconds. Eight times of RA in two minutes. After the FNS treatment, the needle was withdrawn.
  Arms: FSN group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of Fu's Subcutaneous Needling (FSN) in carpal tunnel syndrome (CTS). The main questions it aims to answer are:

* Dose FSN improve the symptoms of CTS?
* Dose FSN decrease cross section area of median nerve in CTS patients?
* Dose FSN have the effect of electrophysiology exam in CTS patients? Participants will receive wrist splinting and FSN treatment respectively. Researchers will compare wrist splinting group with FSN group to see if FSN being effective for CTS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 20-85 years old.
2. Meet the diagnosis of mild to moderate carpal tunnel syndrome.
3. If the patient has carpal tunnel syndrome in both hands, choose the side with mild or moderate carpal tunnel syndrome.
4. After being explained, join the trial voluntarily and sign the subject's consent form.

Exclusion Criteria:

1. Caused by trauma or mass lesion.
2. Thenar muscle atrophy.
3. Electrophysiological examination revealed severe CTS.
4. Chronic kidney disease, rheumatoid arthritis, abnormal thyroid function, diabetes.
5. Psychiatric history or incapable of cooperating with the investigator.
6. Pregnancy.
7. History of substance abuse or long-term steroid use.
8. History of median nerve surgery.
9. Those who do not sign the consent form.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Change of Boston Carpal Tunnel Questionnaire (BCTQ) | Change from baseline at one month after treatment.
  BCTQ
Change of electrophysiology exam | Change from baseline at one month after treatment.
  Exam of motor latency
Change of cross section area of median nerve in ultrasound | Change from baseline at one month after treatment
  cross section area of median nerve

CONTACTS AND LOCATIONS:
Overall Officials: Chih Ying Wu, MD, Study Chair — China Medical University, China
Locations (1):
- China Medical University Hsinchu Hospital, Zhubei, Hsinchu County, Taiwan

IPD SHARING:
Plan to Share IPD: No